CLINICAL TRIAL: NCT00139867
Title: A Multicenter, Open-label Trial to Assess Subject Preference of PARCOPA, Carbidopa/Levodopa Orally Disintegrating Tablets, Compared to Conventional Carbidopa/Levodopa Tablets in Subjects With Stable Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: SP0780
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2014-10-20 (Estimated); Status verified 2009-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

INTERVENTIONS:
Drug: PARCOPA

SUMMARY:
The objective of this trial was to assess subject preference for PARCOPA, carbidopa/levodopa Orally Disintegrating Tablets (ODT), compared with conventional carbidopa/levodopa tablets, in subjects with stable Parkinson's disease.

DETAILED DESCRIPTION:
See approved Package Insert for Adverse Event information.

ELIGIBILITY:
Inclusion Criteria:

* Stable Parkinson's Disease

Exclusion Criteria:

* Not using carbidopa/levodopa tablets

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2004-01; Primary Completion 2004-05 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (1):
- Schwarz, Milwaukee, Wisconsin, United States